CLINICAL TRIAL: NCT07117357
Title: Acute Effects of Neuroathletic Training on Posterior Chain Muscle Strength, Endurance, Proprioception, Dynamic Balance, and Cognitive Performance in Non-Athletic Individuals
Brief Title: Neuroathletic Training Effects on Muscle Strength, Balance, and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, caglar soylu, Associate Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-49
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Neuroathletic Training; Posterior Chain Muscle Strength; Gluteus Maximus; Hamstrings; Erector Spinae Endurance; Proprioception; Cognitive Performance

STUDY DESIGN:
Intervention Model Description: Parallel group design with two arms (experimental and control). Participants are randomly assigned to either the neuroathletic training group or the standard warm-up control group. Each group undergoes a single 20-minute intervention session, with outcomes measured at baseline, immediately post-intervention, 15 minutes post-intervention, and 30 minutes post-intervention. This design allows for direct comparison of the acute effects of neuroathletic training versus a standard warm-up protocol on the specified outcomes.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors, responsible for conducting and analyzing measurements (e.g., muscle strength, balance, proprioception, and cognitive tests), will be blinded to the group allocation of participants to minimize bias in data collection and interpretation. Participants, care providers, and investigators will not be blinded due to the nature of the intervention, which requires active participation and specific instructions for neuroathletic training or standard warm-up protocols.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuroathletic Training (Experimental): Participants will undergo a 20-minute neuroathletic training protocol using the Z-Health® kit, targeting visual, vestibular, and proprioceptive systems. The protocol includes visual reset exercises (eye massage, palming), star chart eye muscle training, saccade training with letter cards, convergence-divergence training, Brock string training, hip and spine extension exercises, saccule activation lunge exercises, slap tap coordination exercises, and pinhole glasses exercises to enhance motor control, balance, and cognitive performance.
  Interventions: Behavioral: Neuroathletic Training Protocol
- Standard Warm-Up (Active Comparator): Participants will perform a 20-minute standard warm-up protocol consisting of 10 minutes of light walking at a moderate pace on flat terrain, followed by 10 minutes of dynamic stretching exercises (10 repetitions each of leg swings, hip flexor stretches, knee hugs, high knees, butt kicks, arm circles, and trunk rotations). This protocol serves as a control to compare against the neuroathletic training intervention.
  Interventions: Behavioral: Standard Warm-Up Protocol

INTERVENTIONS:
Behavioral: Neuroathletic Training Protocol — This intervention involves a 20-minute neuroathletic training session using the Z-Health® kit. It includes visual reset exercises (eye massage, palming), star chart eye muscle training, saccade training with letter cards, convergence-divergence drills using Brock string, vestibular activation through lunges, spinal and hip extension exercises, slap tap coordination drills, and use of pinhole glasses. The aim is to stimulate sensory pathways and enhance neuromotor readiness acutely.
  Other Names: Z-Health®-based neuroathletic training
  Arms: Neuroathletic Training
Behavioral: Standard Warm-Up Protocol — This 20-minute warm-up consists of two components: 10 minutes of light walking at a moderate pace and 10 minutes of dynamic stretching (leg swings, hip flexor stretches, knee hugs, high knees, butt kicks, arm circles, and trunk rotations). It is intended to mimic standard pre-activity routines and serves as the comparator condition.
  Arms: Standard Warm-Up

SUMMARY:
Neuroathletic training is an innovative approach aimed at enhancing neurophysiological processes to improve motor control, reflex responses, balance, proprioception, and cognitive functions. While this method has shown promise in athletes, its acute effects on non-athletic individuals remain underexplored. The posterior chain (gluteus maximus, hamstrings, and erector spinae) plays a critical role in postural stability, movement, and injury prevention. Weakness in these muscles, coupled with poor balance and proprioception, may increase injury risk. Additionally, cognitive performance, including attention and reaction time, is vital for functional activities and may be enhanced through neuroathletic interventions. This study seeks to address the gap in understanding the acute effects of neuroathletic training on non-athletic individuals, providing evidence to support its integration into rehabilitation and injury prevention programs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years.
* No regular physical activity in the past 6 months (IPAQ Short Form: physical activity level >3000 MET-min/week excluded).
* Body Mass Index (BMI) 18.5-24.9 kg/m².
* No history of lower extremity injury or neurological conditions.
* Ability to perform study tests and exercises.
* Written informed consent.

Exclusion Criteria:

* Acute injury in the past 6 months.
* Chronic pain or postural deformities.
* Sensory impairments affecting study participation.
* Musculoskeletal, neurological, respiratory, or cardiovascular conditions limiting exercise.
* History of malignancy.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Gluteus Maximus Muscle Strength (Newton) | Baseline, Immediately Post-Intervention, 15 Minutes Post, 30 Minutes Post
  Assessed using a digital handheld dynamometer (Lafayette Manual Muscle Tester, Model 01165) during maximal voluntary isometric contraction in prone hip extension. Three trials are conducted, and the highest value is recorded.
Erector Spinae Endurance (Seconds) | Baseline, Immediately Post-Intervention, 15 Minutes Post, 30 Minutes Post
  Evaluated using the Biering-Sørensen Test. Participants maintain a horizontal trunk position with the lower body fixed until fatigue. Time is recorded with a stopwatch.
Knee Joint Proprioception (Degrees) | Baseline, Immediately Post-Intervention, 15 Minutes Post, 30 Minutes Post
  Measured using an inclinometer to assess knee joint position sense. Angular deviation from 30° knee flexion target is recorded. The mean error across trials is used as the final score.
Dynamic Balance (Percent Reach Distance) | Baseline, Immediately Post-Intervention, 15 Minutes Post, 30 Minutes Post
  Assessed with the Y-Balance Test in three directions: anterior, posteromedial, and posterolateral. Reach distances are normalized to limb length and averaged to calculate dynamic balance performance.
Cognitive Performance - Stroop Test Reaction Time | Baseline, Immediately Post-Intervention, 15 Minutes Post, 30 Minutes Post
  Assesses selective attention and cognitive interference using the Stroop Color-Word Test. Reaction time is recorded in milliseconds during the incongruent trial phase.
Cognitive Performance - Stroop Test Error Count | Baseline, Immediately Post-Intervention, 15 Minutes Post, 30 Minutes Post
  Assesses accuracy during the Stroop Color-Word Test. The number of errors made during the incongruent trials is recorded.
Cognitive Performance - Trail Making Test Completion Time | Baseline, Immediately Post-Intervention, 15 Minutes Post, 30 Minutes Post
  Assesses visual attention and task-switching using Trail Making Test Parts A and B. Time to complete each part is recorded in seconds.
Cognitive Performance - Trail Making Test Error Count | Baseline, Immediately Post-Intervention, 15 Minutes Post, 30 Minutes Post
  Assesses accuracy during Trail Making Test Parts A and B. The number of errors committed during each test part is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Gulhane Faculty of Physiotherapy and Rehabilitation, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional data protection policies and ethical considerations. The collected data are limited to the scope of the approved protocol and will only be used for internal analysis by the research team.